CLINICAL TRIAL: NCT03189498
Title: A Phase 1, Open-label, Single-dose, Parallel-group Study to Evaluate the Effect of Renal Impairment on the Pharmacokinetics of JNJ-64041575 in Adult Subjects With Various Degrees of Renal Function
Brief Title: A Study to Evaluate the Effect of Renal Impairment on the Pharmacokinetics of JNJ-64041575 in Adult Participants With Various Degrees of Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CR108333; 2017-000875-10 (EudraCT Number); 64041575RSV1006 (Other: Janssen Pharmaceutica N.V., Belgium)
Record Dates: First submitted 2017-06-15; First posted 2017-06-16 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency | interventions — 4'-chloromethyl-2'-deoxy-3',5'-di-O-isobutyryl-2'-fluorocytidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group 1: Participants With Normal Renal Function (Experimental): Adult participants with normal renal function (estimated glomerular filtration rate [eGFR] greater than or equal to [>=] 90 milliliter per minute [mL/min]) will receive a single oral dose of 1,000 milligram (mg) JNJ-64041575 (4*250-mg tablets) on Day 1 of treatment period.
  Interventions: Drug: JNJ-64041575
- Group 2: Participants With Mild Renal Impairment (Experimental): Adult participants with mild impaired renal function (eGFR >=60 to less than [<] 90 mL/min) will receive a single oral dose of 1,000 mg JNJ-64041575 (4*250-mg tablets) on Day 1 of treatment period.
  Interventions: Drug: JNJ-64041575
- Group 3: Participants With Moderate Renal Impairment (Experimental): Adult participants with moderate impaired renal function (eGFR >=30 to <60 mL/min) will receive a single oral dose of 1,000 mg JNJ-64041575 (4*250-mg tablets) on Day 1 of treatment period.
  Interventions: Drug: JNJ-64041575
- Group 4: Participants With Severe Renal Impairment (Experimental): Adult participants with severe impaired renal function (eGFR >= 15 to <30 mL/min) will receive a single oral dose of 1,000 mg JNJ-64041575 (4*250-mg tablets) on Day 1 of treatment period.
  Interventions: Drug: JNJ-64041575
- Group 5: Participants With ESRD With or Without Hemodialysis (Experimental): Adult participants with end-stage renal disease (ESRD) (eGFR <15 mL/min if not on hemodialysis or requiring hemodialysis treatment for at least 3 months before screening if on hemodialysis) will receive a single oral dose of 1,000 mg JNJ-64041575 (4*250-mg tablets) on Day 1 of treatment period. Participants with ESRD on hemodialysis will be dosed on an interdialysis day within 24 hours of their last hemodialysis treatment.
  Interventions: Drug: JNJ-64041575

INTERVENTIONS:
Drug: JNJ-64041575 — All participants will receive a single oral dose of 1,000 mg JNJ-64041575 (4*250 mg tablets) on Day 1.
  Other Names: ALS-008176, lumicitabine

SUMMARY:
The primary purpose of this study is to evaluate the pharmacokinetic (PK) and systemic exposure of JNJ-63549109 and JNJ-64167896 after a single oral dose of JNJ-64041575 in adult participants with various degrees of renal function (mildly, moderately, or severely impaired, or end-stage renal disease [ESRD] with or without hemodialysis) compared to adult participants with normal renal function.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have a body mass index (BMI: body weight in kilogram (kg) divided by the square of height in meters) of 18.0 to 36.0 kilogram per meter square (kg/m^2), extremes included, and a body weight not less than 50.0 kg, inclusive, at screening
* Contraceptive use by female participants, male participants and their female partners should be consistent with local regulations regarding the use of contraceptive methods for participants participating in clinical studies if these are stricter than what is proposed in these inclusion criteria in the protocol

Participants with normal renal function (Group 1):

-Participant must have an estimated glomerular filtration rate (eGFR) >= 90 milliliter per minute (mL/min)

Participants with renal impairment (Groups 2 to 4):

- The following classifications of renal function are used: Mild renal impairment (eGFR greater than or equal to [>=] 60 to less than [<] 90 mL/min), Moderate renal impairment (eGFR >= 30 to <60 mL/min), Severe renal impairment (eGFR >=15 to <30 mL/min)

Participants with end-stage renal disease (ESRD) with or without hemodialysis (Group 5):

* Participant must have an eGFR <15 mL/min if not on hemodialysis
* Participant on hemodialysis treatment must have been on the same hemodialysis regimen for at least 3 months before screening

Exclusion Criteria:

All participants (Groups 1 to 5):

* Participant has any surgical or medical condition that potentially may alter the absorption, metabolism, or excretion of the study drug (example, Crohn's disease), with the exception of renal impairment
* Participant has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (example, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments
* Participant with a history of clinically significant drug allergy such as, but not limited to, sulfonamides and penicillins, or drug allergy diagnosed in previous studies with experimental drugs
* Participant has known allergies, hypersensitivity, or intolerance to JNJ-64041575 or its excipients
* Participants with evidence of an active infection
* Participant is a woman who is pregnant or breastfeeding

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2017-12-06 (Actual); Study Completion 2017-12-06 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Predose, Day 1: 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, and 336 (Day 15) hours postdose
  The Cmax is the maximum observed plasma concentration.
Area Under the Plasma Concentration-time Curve From Time Zero to Last Measurable Concentration (AUC [0-last]) | Predose, Day 1: 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, and 336 (Day 15) hours postdose
  The AUC (0-last) is the area under the plasma concentration-time curve from time zero to the time of the last measurable concentration.
Area Under the Plasma Concentration-time Curve From Time Zero to Infinite Time (AUC [0-infinity]) | Predose, Day 1: 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, and 336 (Day 15) hours postdose
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z); wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.

SECONDARY OUTCOMES:
Number of Participants With Adverse Events as a Measure of Safety and Tolerability | Up to 20 to 28 days after study drug intake (approximately 5 months)
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V., Belgium Clinical Trial, Study Director — Janssen Pharmaceutica N.V., Belgium
Locations (2):
- Germany (2):
  - CRS Clinical Research Services Kiel, Kiel
  - APEX GmbH, München